CLINICAL TRIAL: NCT00931125
Title: Randomized, Double Blinded, Controlled, Two-center Study Assessing the Safety and Efficacy of Intravitreal Ranibizumab as a Preoperative Adjunct Treatment Before Vitrectomy Surgery in Proliferative Diabetic Retinopathy (PDR) Compared to Vitrectomy Alone
Brief Title: Safety and Efficacy of Intravitreal Ranibizumab as a Preoperative Adjunct Treatment Before Vitrectomy Surgery in Proliferative Diabetic Retinopathy (PDR) Compared to Vitrectomy Alone
Acronym: VITARM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Attila Vajas (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor-Investigator, Attila Vajas, MD, University of Debrecen
Organization: University of Debrecen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRFB002AHU03T
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Diabetic Retinopathy
Keywords: Severe proliferative diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Ranibizumab; Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitrectomy with ranibizumab (Active Comparator): Patients receiving adjunct preoperative intravitreal ranibizumab (3±1 days) before vitrectomy surgery
  Interventions: Drug: ranibizumab and vitrectomy
- vitrectomy without ranibizumab (Placebo Comparator): Patients receiving sham treatment before vitrectomy as a comparator arm
  Interventions: Procedure: vitrectomy without preoperative ranibizumab

INTERVENTIONS:
Drug: ranibizumab and vitrectomy — ranibizumab 10mg/ml intravitreal injection, 0,05 ml
  Other Names: Lucentis intravitreal injection.
  Arms: vitrectomy with ranibizumab
Procedure: vitrectomy without preoperative ranibizumab — sham intravitreal injection before vitrectomy surgery
  Arms: vitrectomy without ranibizumab

SUMMARY:
This study investigates the hypothesis that ranibizumab injection given into the eye is a safe, efficacious and helping treatment option applied before surgical intervention of the proliferative diabetic retinal eye disorder.

DETAILED DESCRIPTION:
This is a randomized, double blinded , controlled, two-center study assessing the feasibility, efficacy and safety of intravitreal ranibizumab injection applied as a preoperative adjunct treatment before vitrectomy surgery in severe proliferative diabetic retinopathy (PDR). Comparator arm consists of patients receiving standard vitrectomy alone with sham intravitreal injection preoperatively.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 or older who have signed an informed consent
* Type I or II diabetes mellitus and severe proliferative retinopathy with tractional retinal detachment, tractional-rhegmatogenous retinal detachment, tractional detachment complicated with vitreous haemorrhage or active severe proliferative retinopathy not responding to previous panretinal laser photocoagulation
* study eye BCVA must have at least light perception and must not exceed 70 letters using ETDRS at testing distance 4 meters
* study eye vision decrease must be resulted from severe PDR

Exclusion Criteria:

* Active ocular inflammation or infection
* History of uveitis
* Uncontrolled glaucoma
* High myopia
* Any concurrent intraocular condition in the study eye that in the opinion of the investigator could confound the study results
* Former treatment with anti-angiogenic drugs within 30 days preceding Day 1 in the study eye
* History of vitrectomy within 60 days preceding Day 1 in the study eye
* History of intraocular surgery within 30 days preceding Day 1 in the study eye
* Untreated diabetes mellitus
* Severe hypertension (systolic pressure higher than 160mmHg)
* Current use of systemic medications known to be toxic to the retina
* History of thromboembolic events (incl MI and stroke) within 5 years
* Major surgery within previous 3 months or planned within the next 28 days
* Known coagulation abnormalities or current use of anticoagulative medications other than aspirins
* Known hypersensitivity to ranibizumab or any component of it
* Women of childbearing potential unless 2 methods of birth control applied
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of preoperative intravitreal ranibizumab | OP day
  Efficacy, measured by surgical time, number of intraoperative bleedings, intraoperative retinal breaks,required endodiathermy

SECONDARY OUTCOMES:
Change in BCVA. | 6 months
Effect in anatomical changes. | 3 ±1 days after injection
Safety. | Over 6 months.
Retinal circulation integrity. | Month 1, 3, 6.
  Evaluating the circulation of original retinal vessels, evaluating the size of proliferative vessels (size of leaking areas and number of leaking points measured by Fluorescein angiography )

CONTACTS AND LOCATIONS:
Overall Officials: Attila Vajas, MD, Principal Investigator — National Institute of Pharmacy
Locations (1):
- University of Debrecen, Medical and Health Science Center, Faculty of Medicine, Department of Ophthalmology, Debrecen, Hungary

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074